CLINICAL TRIAL: NCT02497677
Title: Copenhagen Infant Mental Health Project: A Randomized Controlled Trial Comparing Circle of Security-Parenting and Care as Usual as Interventions Targeting Infant Mental Healths Risks
Brief Title: Copenhagen Infant Mental Health Project: Enhancing Parental Sensitivity and Attachment (CIMHP)
Acronym: CIMHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Væver, associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCPH 2015-10
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Infant Social Withdrawal; Maternal Postnatal Depression
Keywords: parental sensitivity; child attachment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circle of Security-Parenting (Experimental): Circle of Security-Parenting (COS-P) is a brief educative group program for parents
  Interventions: Behavioral: Circle of Security -Parenting
- Care as Usual (CAU) (Active Comparator): Care as usual (CAU) i.e. the active control condition will be standard practices for infants and families at risk in Copenhagen.
  Interventions: Behavioral: Care as Usual

INTERVENTIONS:
Behavioral: Circle of Security -Parenting — The COS-P manual and video material has been translated to Danish (Tryghedscirklen - Forældreprogrammet, manual, Lier, 2013). Based on standard video material of parent-infant interactions, parents are trained to see and understand infant attachment behavior and especially to learn about infant miscuing attachment signals. In the current study parents will attend 10 sessions of 1.5 hour duration
  Other Names: COS-P
  Arms: Circle of Security-Parenting
Behavioral: Care as Usual — CAU are different in the three participating districts and vary in content and duration. All three districts offer (a) group interventions for mothers who experience postnatal depressive symptoms and/or (b) extra counselling home-visits by a health nurse. Number and content of extra home-visits vary in accordance with the families' specific needs, and will rarely exceed 12 extra visits per year.
  Other Names: CAU
  Arms: Care as Usual (CAU)

SUMMARY:
Infant mental health is a significant public health issue as early adversity and expose to childhood stress has life-long consequences for the affected children. Helping families at risk correct their adverse effects on the infant has the potential to halt a negative spiral effect where vulnerable parents fail to cope with an at-risk child - which in turn, adds to the child's vulnerability, negatively affects the parents, and so forth. Over a four year period, an estimated 17.600 dyads will be screened in the City of Copenhagen using standardized screening instruments in detecting infant social withdrawal (ADBB) and maternal postnatal depression (EPDS). A sample of 314 eligible parent(s) will enter into a clinical, randomized control trial to test the efficacy of an 8 week group counseling program, Circle of Security Parenting (COS-P) compared to Care as Usual(CAU) in enhancing maternal sensitivity, child attachment and cognitive development. CIMHP is the first large-scale randomized controlled study to test the efficacy of COS-P in promoting parental sensitivity, child attachment and cognitive development in Denmark. Results will provide evidence regarding the efficacy of an American short term indicated parenting group program when implemented in a Scandinavian country.

DETAILED DESCRIPTION:
Background and rationale Infant mental health is a significant public health issue as early adversity and exposure to early childhood stress has life-long consequences for these affected children on outcomes such physical and mental health, educational attainment, labor market success and family formation. Infants are - as a result of their dependency, vulnerability and relative social invisibility - more exposed to mental health risks than older children. Infants may be at risk due to a particular biological risk (e.g. infantile autism, retardation, prematurity, physical disabilities etc) or to psycho-social risks in the family (e.g. mentally ill parents, poverty, drug/alcohol abuse etc). Recent Danish estimates suggest that one in five families is at risk of inadequate parenting resources and child neglect.

There is by now solid evidence that the establishment of attachment relationships, i.e. a stable emotional bond with a caregiver - mostly the parent - is one of the most important developmental milestones in infancy. Early parent-child attachment relationships function as a blueprint for future social relationships and serve as a framework within which children learn how to deal with stressful situations and to regulate the accompanying negative emotions. Insecure and disorganized attachment is a significant risk for longitudinal child development and psychopathology, as the ability to regulate ones feelings of stress and negative emotions is important for a wide range of socio-emotional outcomes ranging from social competence, moral development and empathy, to academic achievement. Recent meta-analyses show that insecure and disorganized children have a higher risk of developing mental problems later in life. Insecurely attached children are also more likely than securely attached children to develop internalizing problems, such as anxiety and depressive symptoms, as well as externalizing problems such as aggressive behavior. For externalizing problems, the risk was even higher for disorganized children. Furthermore, research into early brain development indicates that brain development can be physiologically altered by severe stress imposed by neglect and inadequate parenting during a child's early years.

Evidence from attachment research shows that sensitive parenting, where the parent is alert and able to understand the infant's expression of emotional states and able to manage and meet the infant's needs contingently, adequately and in a comforting way will lead to the establishment of a pattern of secure attachment in the child. Lack of availability, inconsistent availability, misunderstanding of the infant's emotional expression and parental behavior that frightens the infant may all lead to an insure attachment and in the most severe cases a disorganized attachment. This is indicative of a breakdown of an organized (secure or insecure) attachment behavioral strategy. Disorganized attachment is considered to be the result of parental behavior that is frightening for the child. An extreme example of such behavior is child maltreatment, but all sorts of parental behavior that are not comprehensible for the child, such as dissociation, which is common in depressed parents, is potentially frightening for the child. This sort of behavior results in the paradoxical situation that the parent is a source of comfort and a source of fear at the same time. Thus, in stress situations the child does not know what to do, and the behavioral strategy collapses .

Infant social withdrawal indicates infant distress and early attachment disturbances and is a known risk factor for infant mental health. Infant social withdrawal is indicated by a lack of either positive (e.g. smiling, eye contact) or negative vocal protestations. Sustained withdrawal behavior in infants can be seen as a chronic diminution of the attachment system, which is gradually generalized into a diminished engagement and lowered reactivity to the environment at large. In more European countries the use of the validated systematic screening method, Alarm Distress Baby Scale (ADBB) for identifying infant delayed socio-emotional development in infant mental health clinics and in home visiting programs have shown promising results.

Postnatal depression (PND) is another known risk for infant mental health. A meta-analysis shows that up to 19% of new mothers may experience minor or major depression during the first months postpartum. If only including major depression, the prevalence was found to be 7.1 %. In a more recent European study, 1,066 women were followed from pregnancy to 12 months postpartum. The results indicated that 9.6% of new mothers may experience a major depressive episode during the first year after delivery. No estimates were given for minor depression. Most cases develop within the first three months with a peak incidence of about 4-6 weeks.

PND has a substantial impact on the mother, her partner, her family, mother-baby interactions and attachment insecurity and the longer term socio-emotional and cognitive development of the baby, especially when depression occurs in the first year of life. Often, mothers suffering from postnatal depression are emotionally, cognitively and/or behaviorally inhibited or impaired in their ability to recognize and react with appropriate "sensitivity" and "responsiveness" to their children's needs. With regard to the infants of these mothers, higher incidences of negative behaviors, such as social withdrawal, persistent crying, averted gaze or head position, physical neediness and a lack of expression of delight in the presence of their mothers, have been observed. These behaviors increase the mother's experience of stress, which further contributes to the maintenance of maladaptive interactional behavioral patterns. Without improvement in these negative interaction cycles, for example, through early interventions, there is a greater likelihood for infants to develop an insecure-avoidant, an insecure ambivalent or disorganized attachment pattern.

Research on the treatment of women with postnatal depression has shown that treatment that only focuses on the mother (i.e., medication, psychotherapy) is insufficient to buffer against the negative impact of maternal psychopathology on the child's cognitive and psychosocial development, as well as infant-mother attachment quality. Even when depression is effectively treated, this does not seem to "spill over" and improve the mother-infant relationship and long-term infant social-emotional outcomes. Instead, it is necessary to support the depressed mothers in their specific needs in caring and relating to their infants,

Interventions targeting PND delivered in groups have been found to achieve change through the dual process of emotional experience and reflection in an interpersonal context. Group sessions provide a support network, reduce isolation and stigma, provide an environment in which to practice interpersonal and communication skills, shape coping strategies and learn from each other, and enable a number of families to be treated at once. Recently, building on evidence from attachment research, a special focus is given to preventive group programs that enhance parental sensitivity and secure attachment such as the intervention program "Circle of Security (COS)". Based on findings from more studies, COS has proved efficient in enhancing secure attachment as well as reducing maternal depressive symptomatology in high-risk samples, including mothers in prison and mentally ill mothers. The original COS program consists of 20 weekly sessions of 2 hour durations and includes an initial video assessment of parent -child attachment. In the COS intervention graphical illustrations of "the Circle of Security" are used. This Circle is a roadmap that encompasses the three basic control systems; the attachment system, the exploration system and the caregiving system. The parent is illustrated through the pair of hands that hold together the child's world. In COS concepts, "holding" means to serve as a secure base and safe haven. "The top half" of the Circle depicts the child's exploration system and needs. I order to explore, the child needs the parent to serve as a secure base by "watching over," "delighting in," "helping," and "enjoying with" the child. Having a parent that supports exploration helps the child develop his or her own sense of interest, leading to mastery and competency in later years. Along "the bottom half" is the child's attachment needs: "protect me," "comfort me," "delight in me," and "organize my feelings." By delighting in the child, the parent helps the child constructing an internal representation of him- of herself as a loved person and thereby establish self-worth, and by organizing the child's feelings by accepting, sharing and naming them, the parent co-regulates the child's emotions and lays the groundwork of later self-regulation of emotions. The child's needs for comfort and exploration encouragement shift rapidly and the caregiver must continuously adjust to those needs, whenever possible.

Meta-analytic evidence identifies short term group approaches (< 16 sessions), targeting maternal sensitivity as being the most effective, and sensitivity focused interventions conducted with referred at-risk samples (e.g. DSM-III-R depressed mothers), as being more effective than interventions with other groups. Attachment security, in particular, has been found to be readily influenced by sensitivity-focused interventions. The program "Circle of Security Parenting" (COS-P) is a recent and shorter version of COS that consists of eight weekly sessions of two hours durations without the individual video assessment of attachment. In COS-P standard video materials of child attachment behaviors as well as the graphic materials to illustrate the Circle of Security are used. Themes that are covered during the program are: "The Circle of Security", "Exploration of the child's needs in the circle", "Being with your child in the circle", "Exploration of own challenges in meeting child's needs", and "Disruption and repair of the relationship".

To the best of the investigator's knowledge, the effectiveness of COS-P in relation to enhancing maternal sensitivity and the mother-infant relationship has not been fully tested in an RCT design in a general population, making this study the first. Results will provide evidence regarding the efficacy of an American short term indicated parenting group program when implemented in a Scandinavian country. Further, COS-P is a promising approach as health nurses can be trained COS-P therapists in future up-scaling.

ELIGIBILITY:
Inclusion criteria:

* Mother lives in one of the participating three districts of Copenhagen
* Mother is > 18 years old
* Mother has an infant in the age of 2-12 months born at term (Gestational age (GA) 37-42) or born preterm (GA 30-36).
* Mother speaks and understands Danish.
* Mother is screened positive for symptoms of postnatal depression (EPDS >10) and fulfill criteria for diagnosis of depression assessed in a clinical interview (SCID-5/RV) conducted by a psychologist 10-20 days after EPDS screening AND/OR
* Infant is scored to be socially withdrawn in two ADBB assessments (ADBB >5) conducted within a range of 10-20 days when the infant is 2, 4 or 8 months.
* If there is a father/partner this person speaks and understands Danish or English.

Exclusion Criteria:

* Infant autism and/or early retardation
* Maternal bipolar disorder and/or psychotic disorder, known severe intellectual impairment, suicidal ideation and/or recent suicide attempt and/or present alcohol/substance abuse.
* Family intends to move away from the Copenhagen area within the period of the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-07 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | Assessed at follow-up (infant is 12-16 months)
  Maternal sensitivity is observed during five minutes mother-infant interaction (free play), and will be assessed using Coding Interactive behavior (CIB, Feldman, 1998).

SECONDARY OUTCOMES:
Infant-mother attachment quality | Assessed at follow-up (infant is12-16 months)
  Infant-mother attachment will be assessed by the Strange Situation Procedure( Ainswotrth, 1978) is one of the most well-established indicators of how well or poorly toddlers are functioning in their primary attachment relationship (to mother) with long-term consequences for children's social and emotional adaptation throughout childhood and adolescence.
Infant Social withdrawal | Assessed at follow-up (infant is 12-16 months)
  Infant Social Withdrawal will be assessed by the Alarm Distress Baby Scale (ADBB, Guedeney & Fermanian, 2001).
Infants socio-emotional development - maternal and partner's report | Assessed at follow-up (infant is 12-16 months)
  A self-report measure administered to both mother and her partner.
Infant cognitive and language development | Assessed at follow-up (infant is 12-16 months)
  A standardized test situation by a psychologist using the Bayley III Screener (Pearson, 2008)
Maternal Depressive Symptoms | Assessed at follow-up (infant is 12-16 months)
  A self-report measure (EPDS, Cox, Holden & Sagovsky, 1987).
Maternal overall psychological distress | Assessed at follow-up (infant is 12-16 months)
  A self-report measure (SCL-92, Danish version Olsen, Moretnsen & bech, 2004)
Maternal depression diagnosis | Assessed at follow-up (infant is 12-16 months)
  Structural Clinical Interview for DSM-5 Disorders, Research version (First, Williams, Karg & Spitzer, 2015)
Maternal Attachment | Assessed at follow-up (infant is 12-16 months)
  A self-report measure (Experince in Close relationships, ECR, Fraley et al, 2000)
Family Functioning, reported by mother and partner | Assessed at follow-up (infant is 12-16 months)
  A self-report measure (The McMaster Family Functioning Device, FAD, Epstein, Baldwin & Bishop, 1983, Danish version, Thaustum et al, 2009)
Parental Reflective Functioning, reported by mother and partner | Assessed at follow-up (infant is 12-16 months)
  self-report measure (The parental reflective Functioning Questionare, PRFQ-1, Luyten et al, 2009)
Parental Stress, reported by mother and partner | Assessed at follow-up (infant is 12-16 months)
  A self-report measure (The Parenting Stress Index, third edition, PSI, Abidin, 1990, Danish version, Hogrefe Forlag)
Number of extra homes visits by the health nurse | Assessed at follow-up (infant is 12-16 months)
  Reported by the health nurse

CONTACTS AND LOCATIONS:
Overall Officials: Mette Væver, Phd, Principal Investigator — University of Copenhagen
Locations (1):
- UCPH Babylab, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Smith-Nielsen J, Stove LL, Stuart AC, Jakel J, Egmose I, Rohder K, Wendelboe KI, Vaever MS. Differential effects of the circle of security-parenting programme on infant-mother attachment: The role of infant temperament. Br J Clin Psychol. 2025 Dec 18. doi: 10.1111/bjc.70031. Online ahead of print. PMID 41414735
- [Derived] Vaever MS, Smith-Nielsen J, Lange T. Copenhagen infant mental health project: study protocol for a randomized controlled trial comparing circle of security -parenting and care as usual as interventions targeting infant mental health risks. BMC Psychol. 2016 Nov 22;4(1):57. doi: 10.1186/s40359-016-0166-8. PMID 27876079